CLINICAL TRIAL: NCT01388959
Title: Multicentre, Open Label, Phase II Trial to Evaluate the Efficacy and Safety of Treatment With Rituximab in Patients Suffering From Follicular Non-Hodgkin's Lymphoma (FNHL) With Residual Minimal Disease After Autologous Transplantation of hematopoïetic Stem Cell (Bone Marrow or Peripheral Blood)
Brief Title: A Study of MabThera/Rituxan (Rituximab) in Patients With Follicular Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M39012
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]

INTERVENTIONS:
Drug: rituximab [MabThera/Rituxan] — 375 mg/m2 intravenously once a week for 4 weeks

SUMMARY:
This single-arm, open-label, multi-centre study will evaluate the efficacy and safety of MabThera/Rituxan (rituximab) in patients with follicular non-Hodgkin's lymphoma with minimal residual disease after autologous haematopoietic stem cell transplantation (bone marrow or peripheral blood). Two groups of patients will be considered for treatment. Group A: Patients with evaluable minimal tumor mass, Group B: Patients with complete response and abnormal B-cell lymphoma 2 (bcl2) status. Patients will receive MabThera/Rituxan 375 mg/m2 intravenously once every week. The anticipated time on study treatment is 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18-75 years of age
* Diagnosis of follicular non-Hodgkin's lymphoma (FNHL)
* Previously treated with chemotherapy with autologous haemotopoietic stem cell transplantation (bone marrow or peripheral blood cells)

Exclusion Criteria:

* Active viral hepatitis
* Eastern Cooperative Oncology Group (ECOG) performance status >2
* Patients not willing to sign informed consent form

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1998-11; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Treatment response rate according to World Health Organization criteria (Group A) | Day 50
Normalization of B-cell lymphoma 2 levels | Day 50

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | 3 years
Progression-free survival | 3 years
Duration of treatment response | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Toulouse, France